CLINICAL TRIAL: NCT04877756
Title: Phase 2a Prospective, Randomized, Double-blind, Intra-subject, Placebo-controlled, Proof of Concept Study to Evaluate the Efficacy of OLX10010 as an Adjunct Therapy to Reduce the Recurrence of Hypertrophic Scars After Scar Revision Surgery
Brief Title: Study to Evaluate Efficacy of OLX10010 in Reducing Recurrence of Hypertrophic Scarring After Scar Revision Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Olix Pharmaceuticals, Inc. (Industry)
Collaborators: Alira Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: OLX10010-02
Record Dates: First submitted 2021-04-22; First posted 2021-05-07 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Hypertrophic Scar
Keywords: scar revision surgery; OLX10010; siRNA
MeSH Terms: conditions — Cicatrix, Hypertrophic

STUDY DESIGN:
Intervention Model Description: 2 parallel arms and then a 3rd arm will be enrolled if the endpoints for the first 2 arms aren't met.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A 2.0 mg/cm OLX10010 biweekly (Experimental): Arm A- half the scar treated with 2.0 mg/cm of OLX10010 biweekly, other half treated with OLX Placebo
  Interventions: Drug: OLX10010
- Arm B 5.0 mg/cm OLX10010 biweekly (Experimental): Arm B- half the scar treated with 5.0 mg/cm of OLX10010 biweekly, other half treated with OLX Placebo
  Interventions: Drug: OLX10010
- Arm C 2.0 mg/cm OLX10010 weekly (Experimental): Arm C- half the scar treated with 2.0 mg/cm of OLX10010 weekly, other half treated with OLX Placebo
  Interventions: Drug: OLX10010

INTERVENTIONS:
Drug: OLX10010 — Lyophilized cake reconstituted with WFI and injected intradermally
  Other Names: a cell penetrating asymmetric small interference RNA (cp-asiRNA), targeting a gene involved in formation of fibrosis

SUMMARY:
Phase 2a, prospective, randomized, double-blind, intra-subject, placebo-controlled, proof of concept study. Approximately twenty subjects will be randomized 1:1 to one of two treatment arms:

Arm A: 2.0 mg/cm OLX10010 biweekly (every two weeks) Arm B: 5.0 mg/cm OLX10010 biweekly (every two weeks) Each treatment arm will have approximately 10 subjects. Each subject will receive both active (OLX10010) and control (placebo) treatment post-hypertrophic scar surgery biweekly (every two weeks) for a total of six doses. Dosing will occur post-surgery on Weeks 2, 4, 6, 8, 10, and 12. Post-treatment follow-up visits will occur at Weeks 18 and 24, and a long-term follow-up visit will occur at Month 12. The Patient and Observer Scar Assessment Scale (both physician and patient scales), Stony Brook Scar Evaluation Scale, Vancouver Scar Scale, and a photograph-based visual analog scale by blinded experts will be completed prior to scar revision surgery, at Weeks 2, 8, 12, 18, and 24, and at Month 12. The overall opinion responses on the physician scales of the POSAS at Week 24 will be used for primary endpoint analysis.

The total length of the linear hypertrophic scar line will be divided equally for treatment with OLX10010 and placebo, injected intradermally per centimeter (cm). The OLX10010 end and placebo end of the scar line will be separated by a 2 cm or greater distance depending on the scar length.

After the Week 24 visit, all data collected will be cleaned and all data management activities will be completed. After the database is frozen/locked, the primary endpoint efficacy analysis will be completed. If at least one of the treatment arms are shown to be appropriate to reduce recurrence of hypertrophic scars, all analyses will be performed. If the efficacy analysis of Arms A and B indicate the study doses are not as effective as expected, the sponsor may decide to add a third arm (Arm C) to explore the weekly dosing regimen. See detailed summary.

Subjects in all study arms will continue in the study until their Month 12 visit. After all subjects complete that visit, data are collected, and data management activities are completed, Month 12 data will be analyzed.

DETAILED DESCRIPTION:
This is a Phase 2a, prospective, randomized, double-blind, intra-subject, placebo-controlled, proof of concept study. Approximately twenty subjects will be randomized 1:1 to one of two treatment arms:

Arm A: 2.0 mg/cm OLX10010 biweekly (every two weeks) Arm B: 5.0 mg/cm OLX10010 biweekly (every two weeks) Each treatment arm will have approximately 10 subjects. Each subject will receive both active (OLX10010) and control (placebo) treatment post-hypertrophic scar surgery biweekly (every two weeks) for a total of six doses. Dosing will occur post-surgery on Weeks 2, 4, 6, 8, 10, and 12. Post-treatment follow-up visits will occur at Weeks 18 and 24, and a long-term follow-up visit will occur at Month 12. The Patient and Observer Scar Assessment Scale (both physician and patient scales), Stony Brook Scar Evaluation Scale, Vancouver Scar Scale, and a photograph-based visual analog scale by blinded experts will be completed prior to scar revision surgery, at Weeks 2, 8, 12, 18, and 24, and at Month 12. The overall opinion responses on the physician scales of the POSAS at Week 24 will be used for primary endpoint analysis.

The total length of the linear hypertrophic scar line will be divided equally for treatment with OLX10010 and placebo, injected intradermally per centimeter (cm). The OLX10010 end and placebo end of the scar line will be separated by a distance of 2 cm or greater depending on the scar length.

After the Week 24 visit, all data collected will be cleaned and all data management activities will be completed. After the database is frozen/locked, the primary endpoint efficacy analysis will be completed. If at least one of the treatment arms are shown to be appropriate to reduce recurrence of hypertrophic scars, all analyses will be performed. If the efficacy analysis of Arms A and B indicate the study doses are not as effective as expected, the sponsor may decide to add a third arm (Arm C) to explore the weekly dosing regimen:

Arm C: 2.0 mg/cm OLX10010 weekly If added, Arm C will enroll 10 subjects. Each subject will receive both active (OLX10010) and control (placebo) treatment post-hypertrophic scar surgery weekly for a total of 11 doses. Dosing will occur post-surgery on Weeks 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, and 12. Post-treatment follow-up visits will occur on Weeks 18 and 24, and a long-term follow-up visit will occur at Month 12. The Patient and Observer Scar Assessment Scale (both physician and patient scales), Stony Brook Scar Evaluation Scale, Vancouver Scar Scale, and a photograph-based visual analog scale by two blinded independent assessors will be completed prior to scar revision surgery, at Weeks 2, 8, 12, 18, and 24, and at Month 12. The overall opinion responses on the physician scales of the POSAS at Week 24 will be used for primary endpoint analysis. After all subjects in Arm C complete Week 24, all data are collected, and all data management activities are completed, a new database freeze/lock will be performed. Arm C data will be analyzed.

Subjects in all study arms will continue in the study until their Month 12 visit. After all subjects complete that visit, data are collected, and data management activities are completed, Month 12 data will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males or females, aged 18 to 65, inclusive
* Hypertrophic scar in the abdominal region, from previous surgery or injury, present for ≥ 12 months
* Linear hypertrophic scar equal to or greater than 8 cm in length
* Undergoing elective hypertrophic scar revision surgery
* Serum pregnancy test negative for females of childbearing potential
* Males and females of child-bearing potential (e.g., not post-menopausal for at least one year or surgically sterile) must agree to use effective contraception starting at the Screening Visit and continuing until 14 days after the last dose of OLX10010.
* Properly obtained written informed consent

Exclusion Criteria:

* BMI greater than 32 kg/m2. Exceptions to this criteria can be granted for patients just over this value per PI's discretion
* Hypertrophic scars outside the abdominal area, including face, neck, back, limbs, and the thoracic region
* Hypertrophic scar secondary to burns
* Active infection near the scar revision surgery
* Clinically significant wound near the scar revision surgery
* Additional scar(s) within 2 cm of the scar revision surgery
* End-stage renal disease or severe renal impairment as indicated by serum creatinine > 2.5 mg/dL
* Tanning (natural or artificial) within 14 days prior to the screening visit or unwilling to abstain from natural or artificial tanning for four weeks after surgery. Tanning is not recommended for the remainder of the study but will not be an exclusion criteria or reason for early termination.
* Hypertrophic scar treatment within 12 weeks prior to the screening visit, excluding scar revision surgery
* Radiation or chemotherapy within 12 weeks prior to the screening visit
* Treatment with anti-psychotic, anti-cancer, immunosuppressant, or corticosteroids within 12 weeks prior to the screening visit
* Atopic dermatitis, keloid scar, or skin hypersensitivity
* Received elective body sculpting procedures (e.g., CoolSculpting®) for the abdomen within the past 6 months
* Use of tobacco or nicotine-containing products during study participation (Screening Visit through last follow-up visit)
* Female patients who are pregnant or breastfeeding
* Participation in any experimental drug or device study within 30 days prior to the screening visit
* Any clinically significant finding, in the judgement of the treating investigator, that would place the subject at health risk, impact the study, or affect the completion of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2021-08-19 (Actual); Primary Completion 2023-01-11 (Actual); Study Completion 2023-07-12 (Actual)

PRIMARY OUTCOMES:
• Change in recurrence of hypertrophic scar after scar revision surgery measured by physician scar assessment using the overall opinion score on the Observer Scar Assessment Scale at Week 24 | Week 24
  • The change of recurrence of hypertrophic scar will be measured by Observer Scar Assessment Scale to rate Vascularity, pigmentation, thickness, relief, pliability, and surface area on a ten point scale with 1 representing normal sensation or skin and 10 indicating the worst imaginable sensation or skin.

SECONDARY OUTCOMES:
• Change in the recurrence of hypertrophic scar after scar revision surgery measured by patient scar assessment using the overall opinion score on the Patient Scar Assessment Scale at Week 24 | Week 24
  • The change of recurrence of hypertrophic scar will be measured by Patient Scar Assessment Scale to rate Vascularity, pigmentation, thickness, relief, pliability, and surface area on a ten point scale with 1 representing normal sensation or skin and 10 indicating the worst imaginable sensation or skin.
• Recurrence of hypertrophic scar after scar revision surgery at Weeks 2, 8, 12, 18, and 24 and Month 12 according to Physician | Week 24 and Month 12
  • Physician scar assessment: Using Total Observer Score from Observer Scar Assessment Scale which is generated by adding all values rated on the scale for that timepoint. Possible scores will be 6 (normal) up to 60 (worst possible)
• Recurrence of hypertrophic scar after scar revision surgery at Weeks 2, 8, 12, 18, and 24 and Month 12 according to Patient | Week 24 and Month 12
  • Patient scar self-assessment: Using Total Patient Score from Patient Scar Assessment Scale which is generated by adding all values rated on the scale for that timepoint. Possible scores will be 6 (normal) up to 60 (worst possible)
• Scar severity | Week 24 and Month 12
  • Vancouver Scar Scale (VSS) which consists of four variables: vascularity, height (thickness), pliability, and pigmentation. Each variable has four to six possible scores. A total score ranges from 0 to 13, whereby a score of 0 reflects normal skin.
• Assessment of Blinded Photographs by Two Independent Assessors: | Week 24 and Month 12
  The visual analog scale is a photograph-based scale derived from evaluating standardized digital photographs. Two independent assessors, blinded to study arm and timepoint, assess the overall improvement of scar appearance (from 0 as the worst to 10 as the best) by reviewing blinded photographs. Each independent assessor completes the 10 cm VAS for both ends (OLX10010 and placebo) of the scar. Mean values of VAS scores assessed by two independent assessors will be used for efficacy analysis.
• Scar variations | Week 24 and Month 12
  • Stony Brook Scar Evaluation Scale (SBSES) assesses the individual attributes like width, height, color, suture marks, and overall appearance with a binary response (0 or 1) for each. The total score range is from 0 (worst) to 5 (best) scar.
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | Week 24 and Month 12
  • Measured by Adverse Events incidence
Severity of Treatment-Emergent Adverse Events [Safety and Tolerability] | Week 24 and Month 12
  • Measured by Adverse Events severity

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Neumeister, MD, Study Director — OliX Pharmaceuticals
Locations (6):
- United States (6):
  - MedStar Health Research Institute, Washington D.C., District of Columbia
  - Miami Dermatology & Laser Research, LLC, Miami, Florida
  - Miami Plastic Surgery, Miami, Florida
  - Henry Ford Health System, Detroit, Michigan
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Paddington Testing Co, Inc., Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hwang J, Chang C, Kim JH, Oh CT, Lee HN, Lee C, Oh D, Lee C, Kim B, Hong SW, Lee DK. Development of Cell-Penetrating Asymmetric Interfering RNA Targeting Connective Tissue Growth Factor. J Invest Dermatol. 2016 Nov;136(11):2305-2313. doi: 10.1016/j.jid.2016.06.626. Epub 2016 Jul 15. PMID 27427487